CLINICAL TRIAL: NCT03293745
Title: Cognitive Behavioral Therapy for Insomnia: Face-to-Face Versus Telemedicine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: American Academy of Sleep Medicine (Other)
Responsible Party: Principal Investigator, J. Todd Arnedt, Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00130209
Record Dates: First submitted 2017-09-19; First posted 2017-09-26 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Face to Face CBT-I (F2F) (Active Comparator): Participants in the F2F arm will receive a standard 6-session course of Cognitive-Behavioral Therapy for Insomnia (CBT-I) delivered in-person, one-on-one with a qualified and experienced therapist.
  Interventions: Behavioral: Face to Face CBT-I (F2F)
- Telemedicine CBT-I (TM) (Experimental): Participants in the F2F arm will receive a standard 6-session course of Cognitive-Behavioral Therapy for Insomnia (CBT-I) delivered via the American Academy of Sleep Medicine (AASM) Sleep Telemedicine system. This telemedicine system provides an online videoconference platform in which a qualified and experienced therapist will deliver CBT-I to participants who will call in to the video therapy sessions with their provider from their homes using a webcam. All aspects of the treatment will remain identical to standard CBT-I delivered face-to-face, as described above, with the exception that the telemedicine technology will be used to deliver the treatment via video conference.
  Interventions: Behavioral: Telemedicine CBT-I (TM)

INTERVENTIONS:
Behavioral: Face to Face CBT-I (F2F) — CBT-I delivered in-person by the therapist.
  Arms: Face to Face CBT-I (F2F)
Behavioral: Telemedicine CBT-I (TM) — CBT-I delivered via American Academy of Sleep Medicine Telemedicine video conference System by the therapist.
  Arms: Telemedicine CBT-I (TM)

SUMMARY:
The purpose of this study is to compare the effectiveness of Cognitive-Behavioral Therapy (CBT) for insomnia conducted face-to-face with a therapist versus CBT for insomnia conducted using Internet-based videoconference technology.

DETAILED DESCRIPTION:
The objective of this clinical trial is to compare the effectiveness of telemedicine Cognitive-Behavioral Therapy (CBT) for insomnia [via the American Academy of Sleep Medicine Sleep Telemedicine (AASM Sleep TM) platform] to gold standard face-to-face CBT for insomnia. The central hypothesis is that CBT for insomnia delivered by AASM SleepTM will be comparable to face-to-face CBT for insomnia for clinical outcomes and patient satisfaction, but AASM SleepTM will be a more cost effective treatment modality (primarily through reduced costs associated with facility use and patient time). The rationale for the proposed project is rooted in the critical need to disseminate CBT for insomnia using the most effective and efficient modalities, with recognition that therapist involvement likely produces the most favorable outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Current diagnosis of insomnia

Exclusion Criteria:

1. Suspicion of or inadequately treated sleep disorder other than insomnia
2. Presence of psychiatric disorders for which CBT for insomnia may be contraindicated
3. Unstable chronic medical condition directly related to insomnia
4. Routine overnight shift work
5. Previous failed adequate trial of CBT for insomnia
6. Unstable dose of sleep medications
7. Lack of access to reliable WiFi connection in the home

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2019-10-04 (Actual); Study Completion 2019-10-04 (Actual)

PRIMARY OUTCOMES:
Change in Insomnia Severity Index (ISI) | Baseline, post-treatment (about 6 weeks), follow-up (about 12-weeks post-treatment)
  The ISI is a 7-item questionnaire assessing the nature, severity, and impact of sleep problems, with good psychometric properties and sensitivity to change with treatment 0-7 = No clinically significant insomnia 8-14 = Subthreshold insomnia 15-21 = Clinical insomnia (moderate severity) 22-28 = Clinical insomnia (severe)

SECONDARY OUTCOMES:
Client Satisfaction Questionnaire (CSQ-8) | Post-treatment (about 6 weeks)
  The CSQ-8 is an 8-item, easily scored and administered measurement that is designed to measure client satisfaction with services. The items for the CSQ-8 were selected on the basis of ratings by mental health professionals of a number of items that could be related to client satisfaction and by subsequent factor analysis. The CSQ-8 is unidimensional, yielding a homogeneous estimate of general satisfaction with services.
  Scores range from 8 - 32, with high scores indicating greater satisfaction.
Change in Therapy Evaluation Questionnaire (TEQ) | Baseline, post-treatment (about 6 weeks), follow-up (about 12-weeks post-treatment)
  The TEQ is a 7-item scale with 5 questions to assess perceived logic of and confidence in treatment, willingness to repeat treatment, and the likelihood that the treatment will help others and 2 questions assessing therapist warmth and competence.

OTHER OUTCOMES:
Change in Patient Health Questionnaire - 9 (PHQ-9). | Baseline, post-treatment (about 6 weeks), follow-up (about 12-weeks post-treatment)
  The PHQ-9 is a 9-item scale measuring the severity of depressive symptoms (range = 0 - 27, with higher scores reflecting more severe depression).
Change in Generalized Anxiety Disorder Questionnaire - 7 (GAD-7) | Baseline, post-treatment (about 6 weeks), follow-up (about 12-weeks post-treatment)
  The GAD-7 is a 7-item survey that measures the severity of anxiety symptoms (range = 0-21, with higher scores reflecting higher levels of anxiety).
Change in Short-Form Health Survey (SF-12) | Baseline, post-treatment (about 6 weeks), follow-up (about 12-weeks post-treatment)
  The 12-item Short-Form Health Survey (SF-12) is a short-form quality of life measure derived from the Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36), which computes physical and mental composite scale scores ranging from 0 to 100.
Change in Multidimensional Fatigue Inventory (MFI-20) | Baseline, post-treatment (about 6 weeks), follow-up (about 12-weeks post-treatment)
  The MFI-20 is a 20-item scale with five subscales representing dimensions of general fatigue, physical fatigue, mental fatigue, reduced motivation, and reduced activity. Higher scores indicate greater fatigue.
Change in Dysfunctional Beliefs About Sleep Scale (DBAS). | Baseline, post-treatment (about 6 weeks), follow-up (about 12-weeks post-treatment)
  The DBAS is a 16-item measure (range: 0-160, with greater scores reflection greater degrees of negative thinking and beliefs related to sleep which presents a series of negative statements or beliefs about sleep. Patients rate the degree to which they agree with or believe each statement.
Change in Work and Social Adjustment Scale (WSAS). | Baseline, post-treatment (about 6 weeks), follow-up (about 12-weeks post-treatment)
  The WSAS is a 5-item questionnaire assessing perceived degree of impairment in work and social domains. Scores range from 0 to 40, with higher scores reflecting greater levels of impairment.
Change in Cornell Service Utilization Index (CSUI). | Baseline, post-treatment (about 6 weeks), follow-up (about 12-weeks post-treatment)
  The CSUI is a 10-item measure that assesses participants' use of medical and mental health services over a six month period.
Change in Working Alliance Inventory - Short Revised (WAI-SR). | Weekly for about 6 weeks
  The WAI-SR is a 12-item measure that assesses the degree to which patients perceive a positive working relationship with their therapist. Scores range from 12-60, with higher scores reflecting greater levels of perceived working alliance with the therapist.
Change in sleep diary measures | Baseline, daily during the 6-week treatment, post-treatment (about 6 weeks), follow-up (about 12-weeks post-treatment)
  Participants will keep sleep diaries daily for 2 weeks at baseline, during treatment, for 2 weeks post-treatment, and for 2 weeks at 12-week post-treatment follow-up. Primary outcomes will include mean sleep efficiency (SE = total sleep time/time in bed*100)
Change in actigraphy measures | Baseline, post-treatment (about 6 weeks), follow-up (about 12-weeks post-treatment)
  Participants will wear an actigraph for 2 weeks at baseline, for 2 weeks post-treatment and for 2 weeks at 12-week post-treatment follow-up. Outcomes will include mean sleep efficiency (SE = total sleep time/time in bed*100)

CONTACTS AND LOCATIONS:
Overall Officials: Todd Arnedt, PhD, Principal Investigator — University of Michigan Department of Psychiatry
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Arnedt JT, Conroy DA, Mooney A, Furgal A, Sen A, Eisenberg D. Telemedicine versus face-to-face delivery of cognitive behavioral therapy for insomnia: a randomized controlled noninferiority trial. Sleep. 2021 Jan 21;44(1):zsaa136. doi: 10.1093/sleep/zsaa136. PMID 32658298